CLINICAL TRIAL: NCT07108959
Title: Effect of Ultrasound Guided Erector Spinae Plane Block Versus Perioperative Intravenous Lidocaine Infusion on Proinflammatory Cytokines in Breast Cancer Surgeries
Brief Title: ESPB Versus Perioperative Iv Lidocaine Infusion on Proinflammatory Cytokines in Breast Cancer Surgeries
Acronym: ESPB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Abd Elhamid, Assistant Lecturer of Anesthesia and Surgical Intensive Care , Faculty of Medicine, Alexandria University, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0202188
Record Dates: First submitted 2025-06-19; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; ESPB; Lidocaine Infusion
Keywords: breast cancer; ESPB; lidocaine infusion; cytokines
MeSH Terms: conditions — Breast Neoplasms | interventions — Lidocaine; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (Active Comparator): patients will receive ultrasound guided ESPB with 30 ml bupivacaine 0.25%.
  Interventions: Procedure: Erector spinae plane block (Group E)
- Group L (Active Comparator): Patients will receive 1.5mg/kg lidocaine 2%; intravenously as a bolus dose then 1.5mg/kg/hr lidocaine infusion using a 50cc syringe pump intraoperatively.
  Interventions: Procedure: Lidocaine (drug)

INTERVENTIONS:
Procedure: Erector spinae plane block (Group E) — The ultra sound probe will be placed on the paravertebral region in a Sagittal plane about 3 cm lateral to the T5 spinous process on the operating side to locate erector spinae muscle, rhomboid major and trapezius from inward (To reach T5, we used C7 as an anatomical landmark, which is the most prominent vertebrae in the back and count downwards to reach T5. To locate C7, we will use palpation or ultrasound guidance if there is difficulty in palpation). Following visualization of these muscles and the transverse process of T5, the skin will be infiltrated with 5 ml of 2% lidocaine, and then 30 ml bupivacaine 0.25% will be injected in the plane between the erector spinae muscle and transverse process using a 22-G 10-cm nerve block needle.
  Arms: Group E
Procedure: Lidocaine (drug) — Patients in group L will receive an initial bolus of lidocaine 1.5mg /kg over 10 minutes immediately before the induction of general anaesthesia then 1.5mg/kg/hr lidocaine infusion in a 50cc syringe pump intra operatively that will be stopped at the end of surgery.
  Arms: Group L

SUMMARY:
The present study aims to compare the effect of ESPB versus perioperative iv lidocaine infusion on proinflammatory cytokines in breast cancer surgeries.

DETAILED DESCRIPTION:
Breast surgery is a widely performed procedure worldwide, with a significant number of patients experiencing moderate to severe acute pain (30 50%) and developing chronic post-surgical pain (CPSP) (25-68%). CPSP, characterized by persistent or worsening pain in the breast region lasting for at least 3 months after surgery, can have detrimental effects on emotional well being, functional abilities, quality of life, and impose substantial financial burdens on healthcare systems. The pathophysiology of CPSP involves mechanisms such as traumatic nerve injury, neuroinflammation, and central neuronal sensitization. Stress response to cancer surgeries is usually associated with a group of interactions between the endocrinal, the sympathetic, and the immunological systems resulting in imbalance between pro- and anti-inflammatory cytokines in addition to activating an inflammatory cascade. Exaggerated production of inflammatory mediators (e.g. interleukins [ILs] and tumor necrosis factor alpha [TNFα]), and immune cell dysfunction (e.g. CD4 T) can lead to haemodynamic instability or metabolic derangements besides increasing the susceptibility of postoperative infection, resulting in delaying wound healing, multiple organ dysfunction, and postoperative morbidity. Tissue and peripheral nerve injury leads to a local inflammatory reaction accompanied by increased levels of pro-inflammatory cytokines, including interleukin IL-1 and IL-6, which induce peripheral and central nervous system sensitization leading to hyperalgesia. IL-1 induces long-lasting synthesis and release of substance P from peripheral nerve terminals of primary afferent neurons, which may contribute to neurogenic inflammation. The conventional approach to managing postoperative pain relies heavily on opioids, which carries the risk of adverse effects including respiratory depression, addiction, and even mortality. To address these challenges, multimodal analgesic strategies have been proposed to alleviate both acute and chronic postoperative pain following breast surgery. Lidocaine, being used originally as an antiarrhythmic agent, has been found to possess antinociceptive, anti-inflammatory and anti-hyperalgesia properties, making it a potentially useful drug for relieving postoperative pain.

The systemic administration of lidocaine has shown efficacy in relieving neuropathic pain. Previous meta-analyses have demonstrated the effectiveness of intravenous lidocaine in reducing postoperative pain and opioid consumption in patients undergoing spine and abdomen surgery. However, the efficacy of intravenous lidocaine specifically for breast surgery has not been extensively evaluated due to limitations such as small sample sizes and conflicting findings from individual studies. To supply complete analgesia postoperatively for patients undergoing breast surgeries, it is essential to ideally block the dermatomes of the spinal nerves from C5 to T6. Many techniques have been used widely to control pain after breast surgeries as para vertebral block, epidural block, and intercostal block. Although no optimal method has been defined yet, each one of these techniques has some flaws. Epidural block can lead to unwanted block to the opposite side, epidural abscess, epidural haematoma and accidental dural puncture. Paravertebral block can result in an ideal analgesia, but it has drawback that it can be complicated by pneumothorax and it may be difficult to perform. The intercostal nerve block is simple to apply, but it requires to be performed in several segments.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 -60 years.
* Female patients.
* ASA physical status class I - II.
* Elective resectable non metastatic breast cancer.

Exclusion Criteria:

* Patients with history of sensitivity to the studied drugs.
* Patients with cardiac conduction defects.
* Patients with major spine deformities.
* Patients with severe coagulopathy.
* Patients with infection at injection site.
* Patients with preexisting myopathy or neuropathy because it can worsen neurological deficits and increase sensitivity to local anaesthetic toxicity. Additionally, it complicates diagnosis of new symptoms and carries higher medicolegal risk due to difficulty distinguishing anaesthesia effects from disease progression.
* Psychiatric disease or seizure disorder requiring medication within the previous 2 years.
* Opioid tolerant patient.
* Cognitive dysfunction.
* Body Mass Index ( BMI ) more than 35 kg/m2 or less than 18 kg/m2 .

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measuring serum pro-inflammatory cytokines (IL-1, IL-6) levels in pg/ml. | BASELINE, 2 HOURS POSTOPERATIVE AND 24 HOURS POSTOPERATIVE
  by ELISA TECHNIQUE unit pg/ml.

SECONDARY OUTCOMES:
Effect on perioperative Heart rate | 24 hours
  heart rate in beats/min
Effect on perioperative blood pressure | 24 hours
  blood pressure in mmhg
post-operative pain. | 24 hours
  by Visual Analogue Scale ( VAS Scale) score from 0 to 10 , 0 means no pain, 10 means the worst pain
Duration of postoperative analgesia (min). | 24 hours
  time for first rescue analgesia if VAS >4, by Visual Analogue Scale ( VAS Scale) score from 0 to 10 , 0 means no pain, 10 means the worst pain
Perioperative analgesic consumptions. | 24 hours
  intraoperative fentanyl in ug and postoperative morphine mg
Chronic postsurgical neuropathic pain | 3 months
  by Douleur Neuropathique 4 (DN4 score) from 0 to 10, 0 the minimum, 10 the maximum, > 4 means high probability of neuropathic pain
Time to return of bowel function | 24 hours
  time to first pass flatus and to first defecation in hours reported by the patient (physiological parameter)
side effects | 24 hours
  like Bradycardia or tachycardia, hallucination or signs of lidocaine toxicity such as circumoral numbness, tinnitus, anxiety, headache, seizure activity, and arrhythmias.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine , Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
practical and resource barriers